CLINICAL TRIAL: NCT04595019
Title: The HERMES Trial Hypofractionated Expedited Radiotherapy for Men With localisEd proState Cancer. A Phase II Randomised Trial of Ultrahypofractionated Stereotactic Body Radiotherapy in Men With Localised Prostate Cancer
Brief Title: Hypofractionated Expedited Radiotherapy for Men With localisEd proState Cancer
Acronym: HERMES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICR-CTSU/2020/10070; CCR5273 (Other: Sponsor code); 285291 (Other: IRAS ID)
Record Dates: First submitted 2020-07-24; First posted 2020-10-20 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Single centre, randomised phase II trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5 fraction (Active Comparator): MRI-guided radiotherapy, 36.25 Gray (Gy) in 5 fractions (boost to 40 Gy over tumour/prostate CTV) over 10 days.
  Interventions: Radiation: SBRT
- 2 fraction (Experimental): MRI-guided radiotherapy, 24 Gy in 2 fractions (boost to 27 Gy over tumour/prostate CTV) over 8 days.
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — Stereotactic Body Radiotherapy. Ultrahypofractionated radiotherapy.

SUMMARY:
The purpose of this research is to investigate whether stereotactic body radiotherapy (SBRT), precise X-ray treatment, is best given in five treatments (also called fractions) over 10 days or in two treatments over 8 days. SBRT is an accurate way to deliver a high dose of radiotherapy to the prostate in a smaller number of doses. We have considerable experience with 5-dose SBRT and now wish to examine the feasibility and safety of delivering treatment over two, larger, doses. Previous work has shown it is theoretically possible to deliver two fraction SBRT on the MR-linac and previous studies have shown internal radiotherapy (brachytherapy) administered in two fractions to be a safe option for patients with low-risk prostate cancer.

All treatment within this trial will be delivered on a new, state of the art, radiotherapy machine called an MR-linac (Magnetic Resonance Linear Accelerator). It puts together an MRI scanner with a radiotherapy treatment machine called a Linear Accelerator. The use of the MR-linac means there is no extra radiation dose given when taking images (unlike computerized tomography (CT) scans or X-ray), enabling us to adapt the radiotherapy plan each day if needed to more precisely target the prostate. The results of the study will enable us to find out if the new, shorter treatment (2 doses of radiotherapy), has a similar level of side effects as the 5 dose treatment and is suitable for further study.

ELIGIBILITY:
Inclusion Criteria:

1. Men aged ≥18 years
2. Histological confirmation of prostate adenocarcinoma requiring radical radiotherapy
3. Gleason score 3+4 or 4+3 (Grade groups 2 or 3)
4. MRI stage T3a or less
5. PSA <25 ng/ml prior to starting ADT (Androgen deprivation therapy)
6. Patients will be concurrently treated with androgen deprivation therapy (ADT) for at least 6 months, as per standard of care. Men who need longer courses of ADT (maximum 12 months) will be considered on a case-by-case basis, and bicalutamide monotherapy is accepted as an alternative to LHRH (luteinizing hormone-releasing hormone) analogues if required.
7. WHO (World Health Organisation) Performance status 0-2
8. Ability of the participant understand and the willingness to sign a written informed consent form.
9. Ability/willingness to comply with the patient reported outcome questionnaires schedule throughout the study.

Exclusion Criteria:

1. Contraindications to MRI (e.g. pacemaker, potentially mobile metal implant, claustrophobia)
2. International Prostate Symptom Score (IPSS) 13 or higher
3. Post-void residual >100 mls
4. Prostate volume >80cc
5. Comorbidities which predispose to significant toxicity (e.g. inflammatory bowel disease) or preclude long term follow up
6. Unilateral or bilateral total hip replacement, or other pelvic metalwork which causes artefact on diffusion-weighted imaging
7. Previous pelvic radiotherapy
8. Patients needing 2-3 years of ADT due to disease parameters.
9. Previous invasive malignancy within the last 2 years excluding basal or squamous cell carcinomas of the skin, low risk non-muscle invasive bladder cancer (assuming cystoscopic follow up now negative) or small renal masses on surveillance.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-07-29 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Genitourinary (GU) toxicity | 12 weeks
  The proportion of patients experiencing CTCAE (Common Terminology Criteria for Adverse Events) Grade 2+ genitourinary (GU) toxicity from the start of radiotherapy up to 12 weeks post-treatment.

SECONDARY OUTCOMES:
Physician-reported CTCAE Genitourinary (GU) and Gastrointestinal (GI) toxicity | 12 weeks
  Physician-reported CTCAE GU and GI toxicity will be reported during treatment and at 12 weeks post-treatment will be summarised according to grade and treatment received using descriptive statistics at each time point.
Physician-reported CTCAE Genitourinary (GU) and Gastrointestinal (GI) late toxicity | 1, 2 and 5 years
  Late toxicity (CTCAE) at 1, 2 and 5 years post-treatment will be summarised according to grade and treatment received at each time point.
Quality of life patient-reported outcomes | 12 weeks, 1, 2 and 5 years post treatment.
  Combined data from the IPSS (International Prostate Symptom Score), EPIC-26 (Expanded Prostate Index Composite-26), EQ-5D (EuroQol-5D) and IIEF-5 (International Index of Erectile Function) QOL instruments will be summarised. Domain scores from the quality of life patient-reported outcome tools will be derived using standard algorithms with missing data handled accordingly. Domain scores and individual items from the patient questionnaires will be presented graphically at each time point and summarised using descriptive statistics, separately for each treatment group. Changes from baseline will be assessed within treatment groups, and multiple regression models (e.g. ANCOVA, ordinal logistic regression or longitudinal models) will investigate patient and clinical factors that may be associated with change in patient-reported outcomes.
PSA (Prostate Specific Antigen) control and biochemical failure/progression | 2 and 5 years
  Time to event.

OTHER OUTCOMES:
Assess bi-parametric MRI prostate imaging parameters during treatment | 4 and 12 weeks
  Descriptive statistics will be used to report and analyse the change in ADC (Apparent diffusion coefficient) between baseline and 4 weeks and between baseline and 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Tree, BSc, MBBS, FRCR,, Study Chair — Royal Marsden NHS Foundation Trust
Locations (1):
- The Royal Marsden Nhs Foundation Trust, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided